CLINICAL TRIAL: NCT00478374
Title: Transarterial Chemoembolisation With Doxorubicin in Combination With Systemic Administration of Sorafenib for Patients With Hepatocellular Carcinoma
Brief Title: Sorafenib With TACE to Treat Hepatocellular Carcinoma
Acronym: S-TACE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: J-F DUFOUR, University of Bern
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JFD-12581
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Sorafenib; Procedure: Transarterial chemoembolisation with doxorubicin

INTERVENTIONS:
Drug: Sorafenib — Sorafenib 400mg bid
Procedure: Transarterial chemoembolisation with doxorubicin — Transarterial chemoembolisation (TACE)

SUMMARY:
The purpose of this study is to determine the feasibility to combine sorafenib with transarterial chemoembolisation in patients suffering from hepatocellular carcinoma.The hypothesis is that sorafenib may prevent the development and growth of tumoral lesions not treated by chemoembolisation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inoperable HCC, who are candidates for transarterial chemoembolization (TACE).
* Diagnosis of hepatocellular carcinoma based on the EASL's criteria (1).
* Child-Pugh score < 10 (Child A or B),
* Life expectancy superior to 12 weeks at the pre-treatment evaluation.
* Local therapies have been interrupted for at least 4 weeks
* Written informed consent signed
* Age >= 18
* Performance status ECOG 0-1
* Normal organ and marrow function defined as:

  * Haematopoietic: absolute neutrophil count >1,500/mm3, platelet count > 60,000/mm3, haemoglobin > 9g/dL
  * INR < 1.5 ULN and PTT within normal limits
  * Hepatic: AST or ALT < 5 x ULN
  * Renal: creatinine < 1.5 x ULN
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate birth contraception (must be double and methods recorded) prior to study entry and for the duration of the study participation. For both men and women, these adequate birth control measures must be used for at least 3 months after the last administration of study drug.

Exclusion Criteria:

* Active heart disease is defined as congestive heart failure >NYHA (New York Heart Association) class 2; active coronary artery disease (myocardial infarction more than 6 months prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta-blockers or digoxin are permitted) or uncontrolled hypertension.

  * Congestive heart failure, serious cardiac arrhythmia, active coronary artery disease.
  * Thrombotic or embolic events within the past 6 months such as a cerebrovascular accident (including transient ischemic attacks), pulmonary embolism.
  * Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection.
  * Psychiatric illness/social situations that would limit compliance with study requirements.
  * Patients with evidence of active infection will become eligible for reconsideration 7 days after completing antibiotic therapy.
  * HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with sorafenib.
  * Patients who have been treated with sorafenib.
  * Cerebral metastasis.
  * Child-Pugh score C.
  * Hypertension defined as systolic blood pressure greater than 150 mmHg or diastolic pressure greater than 90 mmHg despite optimal medical management.
  * Proteinuria defined as a 24-hour urine protein excretion greater than 1000 mg. Urine dipstick proteinuria of 1+ or greater will require a 24-hour urine to determine eligibility for enrolment.
  * Therapeutic anticoagulation with coumarin, heparins, or heparinoids.
  * Serious non-healing wounds (including wounds healing by secondary intention), acute or non-healing ulcers, or bone fractures within 3 months of fracture.
  * Evidence of bleeding diathesis.
  * Impairment of swallowing that would preclude administration of sorafenib.
  * History of haemoptysis or surgery within the past 28 days.
  * Organ allograft.
  * Pregnant or breastfeeding patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of the administration of sorafenib in patients with hepatocellular carcinoma treated with TACE by determining the MTD. | 2 years

SECONDARY OUTCOMES:
tumor volumetry | 2 years
changes in the blood concentration of tumor marker AFP | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Candinas, Principal Investigator — Inselspital; Markus Borner, Principal Investigator — Inselspital; Jean-François J Dufour, MD, Study Director — Inselspital
Locations (1):
- Inselspital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Result] Dufour JF, Hoppe H, Heim MH, Helbling B, Maurhofer O, Szucs-Farkas Z, Kickuth R, Borner M, Candinas D, Saar B. Continuous administration of sorafenib in combination with transarterial chemoembolization in patients with hepatocellular carcinoma: results of a phase I study. Oncologist. 2010;15(11):1198-204. doi: 10.1634/theoncologist.2010-0180. Epub 2010 Oct 29. PMID 21036880